CLINICAL TRIAL: NCT00005855
Title: A Phase I/II Study to Evaluate the Safety and Tolerance of Escalating Doses of RSR13 Administered With a Fixed Dose of BCNU Every Six Weeks in Patients With Recurrent Malignant Glioma
Brief Title: Efaproxiral Plus Carmustine in Treating Patients With Progressive or Recurrent Malignant Glioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New Approaches to Brain Tumor Therapy Consortium (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067881; NABTT-9806; JHOC-NABTT-9806
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2003-12

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; recurrent adult brain tumor; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Astrocytoma; Oligodendroglioma; Brain Neoplasms; Gliosarcoma | interventions — Carmustine; efaproxiral

INTERVENTIONS:
Drug: carmustine
Drug: efaproxiral

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of efaproxiral when given with carmustine and to see how well they work in treating patients with progressive or recurrent malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the safety and tolerability of escalating doses of efaproxiral (RSR13) when administered concurrently with carmustine in patients with progressive or recurrent malignant glioma.
* Determine the maximum tolerated dose (MTD) of RSR13 when administered with carmustine in this patient population.
* Determine the pharmacokinetic profile of this regimen in these patients.
* Estimate the efficacy of this regimen at the MTD in these patients.

OUTLINE: This is a nonrandomized, open-label, multicenter, dose-escalation study of efaproxiral (RSR13).

Patients receive RSR13 IV over 30 minutes followed 30 minutes later by carmustine IV over 1-2 hours on day 1. Treatment repeats every 6 weeks for a maximum of 6 courses in the absence of unacceptable toxicity or disease progression.

Cohorts of 6-12 patients receive escalating doses of RSR13 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 3 of 6 or 5 of 12 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are accrued to receive treatment with RSR13 and carmustine at the recommended phase II dose.

Patients are followed at 6 weeks and then every 2 months thereafter.

PROJECTED ACCRUAL: A maximum of 48 patients will be accrued for the phase I portion of this study. A maximum of 47 patients will be accrued for the phase II portion of this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant glioma that is progressive or recurrent after radiotherapy with or without chemotherapy

  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
  * Glioblastoma multiforme
* Prior low-grade glioma allowed provided progression has occurred after radiotherapy with or without chemotherapy and then high-grade glioma is found on biopsy
* Measurable disease by serial MRI or CT scan

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Hemoglobin at least 10 g/dL
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* Alkaline phosphatase no greater than 3 times upper limit of normal (ULN)
* SGOT and SGPT no greater than 3 times ULN

Renal:

* Creatinine no greater than 2.0 mg/dL

Pulmonary:

* Resting oxygen saturation on room air at least 90% by pulse oximetry
* FVC, DLCO, and FEV_1 at least 50% of normal

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other serious concurrent medical illness that would preclude study compliance
* No other prior malignancy within the past 5 years except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 3 weeks since prior investigational biologics

Chemotherapy:

* See Disease Characteristics
* No prior nitrosoureas for glioma
* No more than 1 prior chemotherapy regimen
* At least 4 weeks since prior chemotherapy
* No prior efaproxiral

Endocrine therapy:

* Concurrent corticosteroids (e.g., dexamethasone) allowed

Radiotherapy:

* See Disease Characteristics
* At least 90 days since prior radiotherapy

Surgery:

* Not specified

Other:

* At least 3 weeks since other prior investigational drugs or devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2000-07; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability
Maximum tolerated dose
Pharmacokinetic profile
Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Z. New, MD, Study Chair — The University of Texas Health Science Center, Houston
Locations (9):
- United States (9):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas